CLINICAL TRIAL: NCT06357546
Title: Evaluation of the Absence of Intraoperative Bladder Catheterization in Case of Planned Cesarean Section: Multicenter Non-inferiority Randomized Controlled Trial
Brief Title: Evaluation of the Absence of Intraoperative Bladder Catheterization in Case of Planned Cesarean Section
Acronym: C2S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL23_0411; 2023-A02424-41 (Other: N° ID-RCB)
Record Dates: First submitted 2024-03-26; First posted 2024-04-10 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Pregnant Women; Cesarean Section
Keywords: Catheterization Urethral; Cesarean Section; Postpartum Urinary Retention

STUDY DESIGN:
Intervention Model Description: A randomization list by blocks of random size and stratified by center, by scarred uterus (with or without scar) and Body Mass Index (BMI) at the start of pregnancy (<30 and ≥30), will be established by a methodologist independent of the study. Patients will be randomized into each group at a ratio of 1:1.
Who Masked: Care Provider
Masking Description: The care provider carrying out the heterocatheterization will be blinded to the participant's randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Intraoperative bladder catheterization (Active Comparator): Patients will have spontaneous urination in the hour preceding the caesarean section and will have a systematic intraoperative bladder catheterization.
  Interventions: Procedure: Spontaneous urination during the hour before caesarean section.; Procedure: Systematic bladder catherization during caesarean section.
- Arm B: Absence of intraoperative bladder catheterization (Experimental): Patients will have spontaneous urination in the hour preceding the caesarean section but will not have intraoperative bladder catheterization.
  Interventions: Procedure: Spontaneous urination during the hour before caesarean section.

INTERVENTIONS:
Procedure: Spontaneous urination during the hour before caesarean section. — Patients will be asked to urinate by spontaneous urination in the hour before the cesarean section with a cytobacteriological urine examination (ECBU) carried out. An ultrasound check by Bladderscan of the post-void residue will be carried out as soon as the patient will be installed on the intervention table. In the event of post-void residue of more than 150 ml, favoring urinary infections, the patient will be excluded from the research.
Procedure: Systematic bladder catherization during caesarean section. — After implementation of loco-regional analgesia by spinal anesthesia, the patient will be positioned, with a perineal toilet and installation of a bladder catheter type Foley ch. 16.
  Arms: Arm A: Intraoperative bladder catheterization

SUMMARY:
The hypothesis of this trial is that the absence of systematic bladder catheterization in patients performing spontaneous urination in the hour preceding the planned cesarean section under spinal anesthesia would not lead to more bladder heterocatheterization for postpartum urinary retention (RUPP) in the 24 hours post-cesarean section than systematic intraoperative bladder catheterization up to 2 hours post-surgery.

DETAILED DESCRIPTION:
Introduction:

The recommendations for the clinical practice of cesarean section, published by the National College of French Gynecologists and Obstetricians (CNGOF) in 2022, have led to a standardized surgical technique. During this surgery, urinary catheterization is use and allows to avoid urinary retention and give a better chirurgical exposition. But it presents also risks as urinary infection development or pain and discomfort for the patient. Actually, the CNGOF wonders if for women having a cesarean section, preoperative spontaneous urination would reduce urinary complications compared to the placement of an intraoperative bladder catheter. The current literature does not allow to respond satisfactorily to this question. This is why C2S study proposes a cesarean section without urinary catheterization following a spontaneous miction.

Aim:

The aim of this trial is to evaluate the rate of bladder heterocatheterization in cases of postpartum urinary retention (RUPP) within 24 hours following a planned cesarean section under spinal anesthesia, according to two management methods: the absence of intraoperative catheterization associated with spontaneous urination in the hour preceding the cesarean section versus systematic intraoperative bladder catheterization up to 2 hours postoperatively. Moreover, this trial will allows to evaluate benefits and risks of the urinary catheterization absence.

Methods:

Following the aim of the trial, it is a prospective randomized study comparing these two treatment modalities in a randomized controlled study with a high level of evidence.

In order to meet the objectives of the study, 500 patients will be included.

Patients will be informed by the investigator during the Caesarean section scheduling consultation, and included the day before their cesarean section during their hospitalization. They will be randomized by the investigator the day before their cesarean section or on the morning of their cesarean section.

In the hour before the cesarean section, participants will be asked to urinate spontaneously. Once the patient is installed on the operating table, the investigator will carry out an ultrasound check using bladder scan of the post-void residue. In the event of a post-void residue of more than 150 ml, the participant will be removed from the research.

After the surgical closure of the cesarean section (H0) starts the postpartum follow-up.

* Between 2 and 3 hours after H0 (H2-H3), an ultrasound check by bladder scan will be carried out in the recovery room, and after collecting the first spontaneous urination, the urine will be quantified using a graduated cup.
* After the first urination or between 5 and 9 hours after H0 (H5-H9), an ultrasound check of the remaining bladder volume will be carried out by bladder scan.
* No later than H9, a bladder heterocatheterization will be carried out in the following cases:

  * Complete RUPP: absence of spontaneous urination
  * Partial RUPP: volume urinated less than the post-void residue (only if the volume urinated > 150 ml)
* After the first urination or the bladder heterocatheterization, a cyto-bacteriological examination of the urine (ECBU) will be carried out.
* Moreover, the patient will evaluate their pain and discomfort felt during their first urination or heterocatheterization using a visual numerical scale (EVN).
* The clinical team will collect complications and adverse events.
* 24 hours after H0 (H24), a ECBU will be realised and the patient's experience of childbirth will be assessed using the Questionnaire For Assessing the Childbirth Experience (QEVA).
* At H24 and at 6 weeks after the caesarean section (W6), the investigator will collect any additional prescriptions for painkillers.
* From the day of the caesarean section to the last visit at 6 weeks after the surgery, potential adverse events will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient admitted for a planned cesarean section after 34 weeks under spinal anesthesia
* Single or twin pregnancy
* Unscarred or with one or two scars of the uterus

Exclusion Criteria:

* Positive urine test strip showing a presence of nitrites or leukocytes, the day before the surgery suggesting asymptomatic bacteriuria
* Emergency Caesarean
* Scheduled Caesarean section with intervention delayed beyond 3 p.m. for service organization reasons
* Epidural anesthesia
* Contraindication to spinal anesthesia (uncorrected hypovolemia; blood coagulation disorders; sepsis or severe inflammation at the puncture site; neurological deficit; migraine pattern; spinal cord disease; spinal malformation; febrile syndrome)
* ASA (American Society of Anesthesiologists) score ≥ 4
* Placental insertion abnormality (placenta previa and/or accreta)
* Medical indication for monitoring of diuresis
* Oliguria or renal failure
* Indication for use of intrathecal clonidine during scheduled cesarean section
* History of bladder surgery or surgical urological pathology during pregnancy (JJ catheter in place)
* History of complex abdominal surgery
* Impossibility or absence of obtaining free, informed and written consent, after a period of reflection
* Patient not affiliated or beneficiary of a national health insurance system
* Patient under legal protection, under guardianship or under curatorship
* Patient having participated in interventional research on a drug within 3 months before inclusion
* Patient participating in another interventional research
* Patient in exclusion period determined by another study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Necessity of heterocatheterization within 24 hours following the cesarean section. | Between Hour 0 (time of surgical closure) and Hour 24
  Heterocatheterization is indicated in cases of Complete postpartum urinary retention (RUPP-C) or in cases of Partial postpartum urinary retention (RUPP-P) with a post-void residue (measured by Bladder scan) greater than the volume urinated (measured in a graduated jar), provided the volume urinated exceeds 150 ml.

SECONDARY OUTCOMES:
Experience of childbirth | Hour 24
  The participant's experience of childbirth will be assessed using the Questionnaire For Assessing the Childbirth Expérience (QEVA) built in 26 items:
  Score result:
  D1: Emotions during childbirth (Items 1, 2, 3, 4 and 24) D2: Interactions with healthcare professionals (Items 5, 6, 7, 8 and 9) D3: First moments with the child (Items 17, 18 and 19) D4: Delayed emotions (Items 20, 21, 22, 23)
Duration of preoperative preparation | Between entering the surgery room and incision during the surgical procedure
  The duration of preoperative preparation (min) will be measured from entry into the operating room to the incision.
Operating time | During surgery (Between incision and surgical closure)
  Operating time (in minutes) corresponds to the period between incision and surgical closure (H0).
Duration of post-operative hospitalization | Discharge from hospitalization (Maximum 1 month after the cesarean section)
  Duration of post-operative hospitalization (in days and hours) corresponds to the period between surgical closure (H0) and discharge from hospitalization.
Time to resume ambulation | Discharge from hospitalization (Maximum 1 month after the cesarean section)
  The time to resume ambulation (in hours) corresponds to the period between surgical closure (H0) and resumption of ambulation.
First urination | Discharge from hospitalization (Maximum 1 month after the cesarean section)
  The time to the 1st urination (in hours) corresponds to the period between surgical closure (H0) and the 1st urination.
Pain during the first urination or the first heterocatheterization | Between Hours 6 and 9
  The participant will self-assess her pain felt during the first urination or the first heterocatheterization postpartum, using a visual numerical scale (EVN) between 0 to 10 (0 = absence of pain and 10 = maximum pain imaginable), between surgical closure (H0) and 6 hours after (H6) or no later than 9 hours after (H9) in case of urinary retention.
Discomfort during the first urination or the first heterocatheterization | Between Hours 6 and 9
  The participant will self-assess her discomfort felt during the first urination or the first heterocatheterization postpartum, using a visual numerical scale (EVN) between 0 to 10 (0 = absence of discomfort and 10 = major discomfort which can be a burning sensation, pain, etc.), between surgical closure (H0) and 6 hours after (H6) or no later than 9 hours after (H9) in case of urinary retention.
Additional prescription for painkillers | Discharge from hospitalization (Maximum 1 month after the cesarean section)
  The additional prescription for analgesics corresponds to the analgesics necessary postpartum, in addition to basic treatment, and until discharge from hospitalization (Yes or No, and if Yes: Level I, II or III).
Urinary infection detection | Hour 24
  A cyto-bacteriological examination of the urine (CBEU) is realised at the first urination or at the first heterocatheterization postpartum, or 24 hours after surgical closure (H24). The CBEU is positive in case of a bacteriuria ≥ 103 CFU/mL, for Escherichia coli ≥ 104 CFU/mL and for other germs with leukocyturia ≥ 104 CFU/mL.
Occurrence of surgical difficulties | During caesarean section procedure
  The occurrence of surgical difficulties is evaluated by the surgeon during the caesarean section. It can be : bladder distension at the start of the procedure, discomfort during surgical exposure, incision difficulty, uterine splitting line, difficulty in fetal extraction, difficulty in uterine suturing, uterine atony, bladder distension at the end of the procedure, or others.
Occurrence of operative complications | Between surgical incision and discharge of hospitalization (Maximum 1 month after the cesarean section)
  The occurrence of operative complications is evaluated by the surgeon from the start of the intervention (surgical incision) and the discharge of hospitalization. It can be : bladder wound, digestive wound, postpartum hemorrhage defined by bleeding greater than 500 ml within 24 hours after surgical closure, surgical revision, quantity of bleeding in the event of surgical revision, or others.
Amount of bleeding | Between surgical incision and Hour 0, Hour 0 and Hour 3, Hour 3 and Hour 24.
  The measurement of the bleeding quantity (in mL) is done between surgical incision and surgical closure (H0) in the operating room, between H0 and 2 hours after (H2) in recovery room, and between 2 hours (H2) and 24 hours (H24) after surgical closure in hospitalization.
Presence of symptoms suggestive of a urinary infection | Between Hour 24 and the postpartum consultation at 6 weeks +/- 2 weeks
  If the presence of symptoms suggestive of a urinary infection is positive, an authentication of the infection is carried out by CBEU or dipstick. The analysis of this symptoms is done between 24 hours after surgical closure (H24) and the postpartum consultation at 6 weeks +/- 2 weeks.
Presence of functional signs (dysuria, incontinence, delayed bleeding or others) | Between Hour 24 and the postpartum consultation at 6 weeks +/- 2 weeks
  The presence of functional signs (dysuria, incontinence, delayed bleeding or others) is detected between 24 hours between the surgical closure (H24) and the postpartum consultation at 6 weeks +/- 2 weeks.
Time before resuming spontaneous urination | Postpartum consultation at 6 weeks +/- 2 weeks.
  In case of heterocatheterization between surgical closure (H0) and 6 hours after (H6), the time before resuming spontaneous urination is measured (in days) during the postpartum consultation at 6 weeks +/- 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey LAMOUROUX, MD, Study Director — Montpellier University Hospital
Locations (2):
- France (2):
  - Montpellier University Hospital, Montpellier
  - Nîmes University Hospital, Nîmes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sentilhes L, Schmitz T, Madar H, Bouchghoul H, Fuchs F, Garabedian C, Korb D, Nouette-Gaulain K, Pecheux O, Sananes N, Sibiude J, Senat MV, Goffinet F. [The cesarean procedure: Guidelines for clinical practice from the French College of Obstetricians and Gynecologists]. Gynecol Obstet Fertil Senol. 2023 Jan;51(1):7-34. doi: 10.1016/j.gofs.2022.10.002. Epub 2022 Oct 11. French. PMID 36228999
- [Background] Hou D, Jia Y, Han A, Hu Q, Li J, Liang W. Effect of urinary catheter removal at different times after caesarean section: A systematic review and network meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2023 Jan;280:160-167. doi: 10.1016/j.ejogrb.2022.12.002. Epub 2022 Dec 5. PMID 36502759
- [Background] Senanayake H. Elective cesarean section without urethral catheterization. J Obstet Gynaecol Res. 2005 Feb;31(1):32-7. doi: 10.1111/j.1447-0756.2005.00237.x. PMID 15669989
- [Background] Ghoreishi J. Indwelling urinary catheters in cesarean delivery. Int J Gynaecol Obstet. 2003 Dec;83(3):267-70. doi: 10.1016/s0020-7292(03)00144-9. PMID 14643036
- [Background] Acharya S, Uprety DK, Pokharel HP, Amatya R, Rai R. Cesarean section without urethral catheterization: a randomized control trial. Kathmandu Univ Med J (KUMJ). 2012 Apr-Jun;10(38):18-22. doi: 10.3126/kumj.v10i2.7337. PMID 23132469
- [Background] Pandey D, Mehta S, Grover A, Goel N. Indwelling Catheterization in Caesarean Section: Time To Retire It! J Clin Diagn Res. 2015 Sep;9(9):QC01-4. doi: 10.7860/JCDR/2015/13495.6415. Epub 2015 Sep 1. PMID 26500959
- [Background] Abdel-Aleem H, Aboelnasr MF, Jayousi TM, Habib FA. Indwelling bladder catheterisation as part of intraoperative and postoperative care for caesarean section. Cochrane Database Syst Rev. 2014 Apr 11;2014(4):CD010322. doi: 10.1002/14651858.CD010322.pub2. PMID 24729285
- [Background] Li L, Wen J, Wang L, Li YP, Li Y. Is routine indwelling catheterisation of the bladder for caesarean section necessary? A systematic review. BJOG. 2011 Mar;118(4):400-9. doi: 10.1111/j.1471-0528.2010.02802.x. Epub 2010 Dec 23. PMID 21176084
- [Background] Fuchs F, Benhamou D. [Post-partum management after cesarean delivery. Guidelines for clinical practice]. J Gynecol Obstet Biol Reprod (Paris). 2015 Dec;44(10):1111-7. doi: 10.1016/j.jgyn.2015.09.020. Epub 2015 Oct 31. French. PMID 26527019
- [Background] Wei G, Harley F, O'Callaghan M, Adshead J, Hennessey D, Kinnear N. Systematic review of urological injury during caesarean section and hysterectomy. Int Urogynecol J. 2023 Feb;34(2):371-389. doi: 10.1007/s00192-022-05339-7. Epub 2022 Oct 17. PMID 36251061
- [Background] Bartzen PJ, Hafferty FW. Pelvic laparotomy without an indwelling catheter. A retrospective review of 949 cases. Am J Obstet Gynecol. 1987 Jun;156(6):1426-32. doi: 10.1016/0002-9378(87)90012-3. PMID 3591859
- [Background] Sentilhes L, Vayssiere C, Deneux-Tharaux C, Aya AG, Bayoumeu F, Bonnet MP, Djoudi R, Dolley P, Dreyfus M, Ducroux-Schouwey C, Dupont C, Francois A, Gallot D, Haumonte JB, Huissoud C, Kayem G, Keita H, Langer B, Mignon A, Morel O, Parant O, Pelage JP, Phan E, Rossignol M, Tessier V, Mercier FJ, Goffinet F. Postpartum hemorrhage: guidelines for clinical practice from the French College of Gynaecologists and Obstetricians (CNGOF): in collaboration with the French Society of Anesthesiology and Intensive Care (SFAR). Eur J Obstet Gynecol Reprod Biol. 2016 Mar;198:12-21. doi: 10.1016/j.ejogrb.2015.12.012. Epub 2015 Dec 21. PMID 26773243
- [Background] Vincent A, Ayzac L, Girard R, Caillat-Vallet E, Chapuis C, Depaix F, Dumas AM, Gignoux C, Haond C, Lafarge-Leboucher J, Launay C, Tissot-Guerraz F, Fabry J; Mater Sud-Est Study Group. Downward trends in surgical site and urinary tract infections after cesarean delivery in a French surveillance network, 1997-2003. Infect Control Hosp Epidemiol. 2008 Mar;29(3):227-33. doi: 10.1086/527512. PMID 18257692
- [Background] Yip SK, Sahota D, Chang AM. Determining the reliability of ultrasound measurements and the validity of the formulae for ultrasound estimation of postvoid residual bladder volume in postpartum women. Neurourol Urodyn. 2003;22(3):255-60. doi: 10.1002/nau.10112. PMID 12707878
- [Background] Demaria F, Amar N, Biau D, Fritel X, Porcher R, Amarenco G, Madelenat P, Benifla JL. Prospective 3D ultrasonographic evaluation of immediate postpartum urine retention volume in 100 women who delivered vaginally. Int Urogynecol J Pelvic Floor Dysfunct. 2004 Jul-Aug;15(4):281-5. doi: 10.1007/s00192-004-1159-3. PMID 15517675
- [Background] Laterza RM, Sievert KD, de Ridder D, Vierhout ME, Haab F, Cardozo L, van Kerrebroeck P, Cruz F, Kelleher C, Chapple C, Espuna-Pons M, Koelbl H. Bladder function after radical hysterectomy for cervical cancer. Neurourol Urodyn. 2015 Apr;34(4):309-15. doi: 10.1002/nau.22570. Epub 2014 Feb 12. PMID 24519734
- [Background] Lim JL. Post-partum voiding dysfunction and urinary retention. Aust N Z J Obstet Gynaecol. 2010 Dec;50(6):502-5. doi: 10.1111/j.1479-828X.2010.01237.x. Epub 2010 Nov 2. PMID 21133858
- [Background] de Boer HD, Detriche O, Forget P. Opioid-related side effects: Postoperative ileus, urinary retention, nausea and vomiting, and shivering. A review of the literature. Best Pract Res Clin Anaesthesiol. 2017 Dec;31(4):499-504. doi: 10.1016/j.bpa.2017.07.002. Epub 2017 Jul 8. PMID 29739538
- [Background] Hernandez NS, Wang AY, Kanter M, Olmos M, Ahsan T, Liu P, Balonov K, Riesenburger RI, Kryzanski J. Assessing the impact of spinal versus general anesthesia on postoperative urinary retention in elective spinal surgery patients. Clin Neurol Neurosurg. 2022 Nov;222:107454. doi: 10.1016/j.clineuro.2022.107454. Epub 2022 Sep 27. PMID 36201900
- [Background] Baldini G, Bagry H, Aprikian A, Carli F. Postoperative urinary retention: anesthetic and perioperative considerations. Anesthesiology. 2009 May;110(5):1139-57. doi: 10.1097/ALN.0b013e31819f7aea. PMID 19352147
- [Background] Neron M, Fatton B, Monforte M, Mares P, de Tayrac R, Letouzey V. [Evaluation of urine postvoid residuals in post-partum period: a prospective and descriptive clinical study]. Prog Urol. 2015 Mar;25(4):211-6. doi: 10.1016/j.purol.2014.09.043. Epub 2014 Oct 22. French. PMID 25450754
- [Background] Neron M, Allegre L, Huberlant S, Mousty E, de Tayrac R, Fatton B, Letouzey V. Impact of systematic urinary catheterization protocol in delivery room on covert postpartum urinary retention: a before-after study. Sci Rep. 2017 Dec 18;7(1):17720. doi: 10.1038/s41598-017-18065-8. PMID 29255204
- [Background] Nasr AM, ElBigawy AF, Abdelamid AE, Al-Khulaidi S, Al-Inany HG, Sayed EH. Evaluation of the use vs nonuse of urinary catheterization during cesarean delivery: a prospective, multicenter, randomized controlled trial. J Perinatol. 2009 Jun;29(6):416-21. doi: 10.1038/jp.2009.4. Epub 2009 Feb 12. PMID 19212327
- [Background] Basbug A, Yuksel A, Ellibes Kaya A. Early versus delayed removal of indwelling catheters in patients after elective cesarean section: a prospective randomized trial. J Matern Fetal Neonatal Med. 2020 Jan;33(1):68-72. doi: 10.1080/14767058.2018.1487394. Epub 2018 Jul 18. PMID 29886771
- See also: National perinatal survey: Births, two-month follow-up and establishments - Situation and evolution since 2016 — http://enp.inserm.fr/wp-content/uploads/2023/09/ENP2021_Rapport_MAJ_Juin2023.pdf
- See also: Birth rate - Fertility - Tables of the French economy | Insee — http://www.insee.fr/fr/statistiques/4277635?sommaire=4318291
- See also: Analysis and improvement of practices: planned cesarean sections at term — http://www.has-sante.fr/upload/docs/application/pdf/2016-10/cesariennes_programmees_a_terme_rapport_long.pdf
- See also: What are the main principles of RAC for planned cesarean section? — http://www.youtube.com/@pedagogienumeriqueensante314/search?query=fuchs